CLINICAL TRIAL: NCT06710873
Title: Analysis of Clinical Application of China's First Batch of TYRX Absorbable Antibacterial Envelope
Status: Active, not recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2024-911-01
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-11

CONDITIONS: CIED Infection; TYRX Absorbable Antibacterial Envelope

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: TYRX Absorbable Antibacterial Envelope — All enrolled patients will receive the TYRX Absorbable Antibacterial Envelope implanted simultaneously during the CIED surgery.

SUMMARY:
This study is the first to use TYRX domesticly, reporting and summarizing its usage to validate its real-world effectiveness in CIED infection prevention.

DETAILED DESCRIPTION:
This study is the first to use TYRX domesticly, reporting and summarizing its usage to validate its real-world effectiveness in CIED infection prevention.

ELIGIBILITY:
Inclusion Criteria:

* All patients who received the TYRX absorbable antimicrobial envelopes at our hospital from December 2023 to September 2024

Exclusion Criteria:

* Allergies to the envelope materials or antimicrobial drugs (minocycline and other tetracyclines, rifampin)
* Existing infections at the CIED implantation site
* Pregnant or breastfeeding women
* children and adolescents

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients who received the TYRX absorbable antimicrobial envelopes at our hospital from December 2023 to September 2024
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
CIED infection | three months post-surgery
  The infection rate related to CIEDs at three months post-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Sun-Yatsen Memorial Hospital of Sun-Yatsen University, Guangzhou, Guangdong, China